CLINICAL TRIAL: NCT04837781
Title: The Effect of Vitamin D3 on the Rate of Orthodontic Tooth Movement (Conventional and Accelerated): Clinical Trial
Brief Title: The Effect of Vitamin D3 on the Rate of Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mushriq F. Abid, Assistant Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178420
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Tooth Position Anomalies
Keywords: Orthodontic, tooth movement, acceleration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding to treatment allocation was possible only for the investigator and data analyst because the clinicians could know the intervention as osteo-perforation can be obviously seen clearly. Masking the intervention for the participants were not possible because micro-osteoperforation is a surgical procedure. All the trial documents were labeled with the study ID number, which was used for participant identification and data collection without unmasking the allocation group. This allowed the investigator to complete data collection and measurements blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal vitamin D (Experimental): Include patients with normal vitamin D level (above 30ng/ml). Vitamin D level will be measured at the beginning of treatment if there is deficiency then the patient refer to specialized physician to be supplied with vitamin D supplement to optimized the level to normal then start orthodontic treatment
  Interventions: Procedure: Micro-osteoperforation
- Vitamin D deficiency (Experimental): Include patients with unknown vitamin D level until time of canine retraction where we measure level if deficiency exist (below 30ng/ml) then the patient will be referred to specialized physician to be supplied with vitamin D supplement.
  Interventions: Procedure: Micro-osteoperforation
- Control (Experimental): includes patients with unknown vitamin D level until the completion of canine retraction where we measure level. If deficiency exists (below 30ng/ml) then we will refer the patient to specialized physician to be supplied with vitamin D supplement
  Interventions: Procedure: Micro-osteoperforation

INTERVENTIONS:
Procedure: Micro-osteoperforation — Micro-osteoperforation Mini-implant facilitated micro-osteoperforation (MOPs) were placed in the experimental side before canine retraction. Three MOPs were placed distal to canine on experimental sides in all group.
  Other Names: MOP

SUMMARY:
The aim of this study is to evaluate the effect of vitamin D3 deficiency on the rate of orthodontic tooth movement in both conventional and accelerated orthodontic. Assessing both lower anterior teeth alignment and the rate of maxillary canine retraction.

DETAILED DESCRIPTION:
To evaluate the effect of vitamin D deficiency on the rate of orthodontic tooth movement in both conventional and accelerated orthodontic, additionally find the effect of vitamin D deficiency on molar anchorage loss, canine rotation, lower incisor crowding alignment time, pain experienced by the patient during OTM and rate of orthodontically induce apical root resorption.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 to 30 years, from both sex.
2. Healthy general medical condition, healthy periodontal condition.
3. Malocclusion that requires extraction of the maxillary first premolars, followed by canine retraction, with moderate lower incisor crowding (Little's irregularity index 3-6mm).
4. Normal shape and structure of maxillary canine, with no history of filling or root canal treatment and normal shape and structure of maxillary first molar.

Exclusion Criteria:

1. Pregnant women.
2. Patient with renal or liver disease.
3. Patient taking corticosteroid or anticonvulsant drugs.
4. Patient with thyroid or parathyroid problems.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-23 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Canine retraction rate | 4 weeks
  Maxillary study model will be 3D scan using optical 3D scanner(Smart Optic,Germany) then measurement done on digital model using 3D program( DentalCad,Galway,3.0,2021),to measure distance from tip of canine to 3rd palatal raguea on both side
Canine retraction rate | 8 weeks
  Maxillary study model will be 3D scan using optical 3D scanner(Smart Optic,Germany) then measurement done on digital model using 3D program( DentalCad,Galway,3.0,2021),to measure distance from tip of canine to 3rd palatal raguea on both side
Canine retraction rate | 12 weeks
  Maxillary study model will be 3D scan using optical 3D scanner(Smart Optic,Germany) then measurement done on digital model using 3D program( DentalCad,Galway,3.0,2021),to measure distance from tip of canine to 3rd palatal raguea on both side
Canine retraction rate | 16 weeks
  Maxillary study model will be 3D scan using optical 3D scanner(Smart Optic,Germany) then measurement done on digital model using 3D program( DentalCad,Galway,3.0,2021),to measure distance from tip of canine to 3rd palatal raguea on both side

SECONDARY OUTCOMES:
Alignment efficiency | 4 weeks
  3D scanned study models were used to measure the amount of crowding in the mandibular anterior teeth using 3Dprogram (DentalCad,Galway,3.0,2021). If Little's irregularity index is less than 1mm and alignment improvement not above 0.5 mm between two successive visits, then treatment is regarded as finished.
Alignment efficiency | 8 weeks
  3D scanned study models were used to measure the amount of crowding in the mandibular anterior teeth using 3Dprogram (DentalCad,Galway,3.0,2021). If Little's irregularity index is less than 1mm and alignment improvement not above 0.5 mm between two successive visits, then treatment is regarded as finished.
Alignment efficiency | 12 weeks
  3D scanned study models were used to measure the amount of crowding in the mandibular anterior teeth using 3Dprogram (DentalCad,Galway,3.0,2021). If Little's irregularity index is less than 1mm and alignment improvement not above 0.5 mm between two successive visits, then treatment is regarded as finished.
Root resorption | 12 weeks
  The amount of root resorption was measured at the start of treatment and after 12 weeks, the length of the root was recoded at these time intervals. Radiographic films were positioned using a customized sensor holder for the lower anterior teeth with a 7cm film-cone distance using long cone paralleling technique. The radiographs were made at 70kV and 8mA DC with an exposure of 0.25 seconds.
pain perception | 7 days
  Evaluations of pain/discomfort was made in the evening on a daily basis over the first 7 days after bonding using a 10- point visual analog scale (VAS) of 10cm length. The highest pain level experienced should be reported by each patient.
  The recording sheet was received by all the patients on the day of bonding, it included seven visual analog scales (one for each day) and the patients were given oral instructions on how to finish the VAS by marking the point on the line which supposed to represent the maximum pain that they felt per day, with 0 refers to "no pain" and 10 refers to "intolerable pain". Patients were reminded daily by a phone call or a text message to mark the recording sheet and to bring it on their next appointment

CONTACTS AND LOCATIONS:
Overall Officials: Mushriq Abid, MSc, PhD, Principal Investigator — University of Baghdad
Locations (1):
- College of Dentisry-University of Baghdad, Baghdad, Al-Rusafa, Iraq

REFERENCES:
- [Derived] Al-Attar A, Abid M. The Effect of Vitamin D3 on the Alignment of Mandibular Anterior Teeth: A Randomized Controlled Clinical Trial. Int J Dent. 2022 Feb 14;2022:6555883. doi: 10.1155/2022/6555883. eCollection 2022. PMID 35198025